CLINICAL TRIAL: NCT02650050
Title: Micropulsed Laser in Association With Intravitreal Injections of Anti-VEGF for the Treatment of Macular Edema in Diabetic Patients (LAMED).
Brief Title: Micropulsed Laser in Association With Anti-VEGF for the Treatment of Macular Edema in Diabetic Patients (LAMED).
Acronym: LAMED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Number of eligible patients too low
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO_2015_28
Record Dates: First submitted 2016-01-07; First posted 2016-01-08 (Estimated); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Macular Edema; Mellitus Diabetes
MeSH Terms: conditions — Macular Edema; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Micropulsed laser photocoagulation (Experimental)
  Interventions: Radiation: Micropulsed laser photocoagulation
- Sham micropulsed laser photocoagulation (Sham Comparator)
  Interventions: Radiation: Micropulsed laser photocoagulation

INTERVENTIONS:
Radiation: Micropulsed laser photocoagulation — Micropulsed laser photocoagulation after 3 anti-VEGF injections

SUMMARY:
Diabetes is a major cause of blindness in adults in the developed countries. The retinal damages associated with diabetes lead to gradual loss of vision, which is accentuated when the macula is affected. This results in macular edema.

Currently, intravitreal injections of anti-VEGF have demonstrated their effectiveness and are the first line treatment of macular edema.

Subthreshold micropulsed laser photocoagulation is an alternative to conventional grid photocoagulation. By delivering pulsed impacts under the thermal lesion threshold of the pigment epithelium, it would not cause the side effects of conventional photocoagulation. Micropulsed photocoagulation combined to anti-VEGF injections, could be the most effective treatment with a minimum injection number and without epithelial lesions.

The main objective of this study is to show that the subthreshold micropulsed laser photocoagulation, in association with intravitreal injections of anti-VEGF, allows to reduce the number of anti-VEGF injections during the first year of treatment.

In this randomized, double blind study, eligible patients will be randomized between a micropulsed laser photocoagulation arm and a sham micropulsed laser photocoagulation arm.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or more
* macular edema associated with a 1 or type 2 diabetes with a hemoglobin A1C level over 5.5% and under <13%
* indication for a treatment with intra-vitreal injections of ranibizumab

Exclusion Criteria:

* treatment with anti-VEGF during the previous 2 months
* treatment by intra-vitreous implant of dexamethasone during the previous six months
* previous history of vitrectomy or glaucoma
* photocoagulation during the previous 3 months
* patient's opposition to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-01-19 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2019-06-04 (Actual)

PRIMARY OUTCOMES:
Number of intra-vitreal anti-VEGF injections | One year

SECONDARY OUTCOMES:
Time to reduction of the macular thickness | One year

CONTACTS AND LOCATIONS:
Overall Officials: Georges CAPUTO, Principal Investigator — Fondation ophtalmologique de Rothschild
Locations (1):
- Fondation ophtalmique Adolphe de Rothschild, Paris, France